CLINICAL TRIAL: NCT02154724
Title: Clinical Investigation for Adaptive Deep Brain Stimulation (aDBS)Closed-loop Device Controlled by Local Field Potentials in Parkinson's Disease.
Brief Title: Clinical Study for Adaptive Deep Brain Stimulation (aDBS)Controlled by Intracerebral Activity in Parkinson's Disease
Acronym: ADBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ADBS-2013-IRCCSMaggioreH
Record Dates: First submitted 2014-05-19; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Parkinson's Disease
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- aDBS (Other): The aDBS (adaptive Deep Brain Stimulation) device is applied both in aDBS and in DBS modality, for two hours in random order for two days. The aDBS can be programmed to deliver aDBS controlled by local fields potential or conventional DBS.
  Interventions: Device: aDBS; Device: DBS

INTERVENTIONS:
Device: aDBS — The aDBS is applied for 2 hours for two days with two different modalities (aDBS and DBS) in random order.
  Other Names: adaptive deep brain stimulation; Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico
Device: DBS — The aDBS s applied for two hous in DBS modality.
  Other Names: Deep Brain Stimulation; Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico

SUMMARY:
Despite its therapeutic effectiveness in Parkinson's disease (PD) the current deep brain stimulation (DBS) strategy could achieve an even better clinical result by adapting to patient's condition. As intracerebral activity analyzed by recording local field potentials (LFPs) from DBS electrodes correlates to PD symptoms, a new stimulation approach would be an "intelligent" adaptive DBS system able to change stimulation settings automatically to the patient's needs using LFPs as control variable.

DETAILED DESCRIPTION:
Despite their proven efficacy in treating Parkinson's disease (PD), deep brain stimulation (DBS) systems could be further optimized to maximize treatment benefits. In particular, because current DBS strategies based on fixed stimulation settings leave the typical parkinsonian motor fluctuations and rapid symptom variations partly uncontrolled, research has focused on developing a novel adaptive DBS (aDBS) system able to adapt moment-by-moment to the patient's clinical condition. aDBS consists of a simple closed-loop model designed to measure and analyze a control variable reflecting the patient's clinical condition to change stimulation settings and send them to an "intelligent" implanted stimulator.

Intracerebral activity analyzed by recording local field potentials (LFPs) from electrodes implanted for DBS in the past 15 years has helped in clarifying basal ganglia pathophysiology and its relation to PD symptoms. Many LFP studies have revealed unknown functions of basal ganglia in PD patients during the execution of motor, cognitive, and behavioral task showing the existence of a "code" in LFP oscillations corresponding to the of patient's clinical condition. LFP-clinical correlations should provide the rationale for developing and implementing new aDBS devices able to adapt stimulation parameters moment-by-moment to the individual patient's needs using LFPs as a control variable for feedback.

ELIGIBILITY:
Inclusion Criteria:

Each patient affected by Parkinson's Disease and implanted with DBS electrodes, following the inclusion criteria of L.I.M.P.E., 2003

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of improvement in unified parkindon's disease rating scale (UPDRS score) of aDSB compare to cDBS | up to1 year
Number of participants with adverse events | up to 1 year
  Counting the number of patient with adverse events (adimensional unit)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Milano, Italy